CLINICAL TRIAL: NCT05917262
Title: Comparing Preoperative Mindfulness-based Breath Training and Heart Rate Variability Biofeedback for Shoulder Surgery Patients in the Postoperative Pain, Shoulder Function, Emotion, Sleep, Quality of Life, Cognitive Function, and Electroencephalography
Brief Title: Comparing Mindfulness-based Breath Training and Heart Rate Variability Biofeedback for Shoulder Surgery Patients in the Postoperative Pain.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Poyu Chen, Assistant professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202202303B0
Record Dates: First submitted 2023-05-17; First posted 2023-06-23 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative; Shoulder Pain
Keywords: Shoulder pain; Postoperative pain; mindfulness; HRV; biofeedback
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-based breathing (Experimental): 20-minute mindfulness-based breathing training
  Interventions: Behavioral: Mindfulness-based breathing
- HRV biofeedback (Experimental): 20-minute HRV biofeedback
  Interventions: Behavioral: HRV biofeedback
- cognitive-behavioral pain psychoeducation (Active Comparator): 20-minute psychoeducation session
  Interventions: Behavioral: cognitive-behavioral pain psychoeducation

INTERVENTIONS:
Behavioral: Mindfulness-based breathing — The 20-minute mindfulness session is a scripted mindfulness exercise that incorporates mindfulness principles of intentionally paying attention to present-moment experiences in a non-judgmental fashion.
  Arms: Mindfulness-based breathing
Behavioral: HRV biofeedback — The 20-minute HRV biofeedback is based on the resonant frequency breathing with an external pacemaker. Generally, the breath rhythm is between 4.5 and 6.5 times per min.
  Arms: HRV biofeedback
Behavioral: cognitive-behavioral pain psychoeducation — The 20-minute psychoeducation session is a supportive session where behavioral coping strategies for pain management are discussed.
  Arms: cognitive-behavioral pain psychoeducation

SUMMARY:
Although shoulder surgeries can effectively relieve pain intensity and restore shoulder function, some patients reported persistent post-operative pain at the 6-month post-surgery follow-up visit. This randomized study aims to determine the effectiveness of three different types of bio-psychosocial support to pre-operative shoulder surgery patients. This study will examine the differential effects of brief mindfulness-based breathing, heart rate variability biofeedback (HRV-BF), and cognitive behavioral pain psychoeducation for pre-operative patients.

ELIGIBILITY:
Inclusion Criteria:

shoulder pain patients with

* (1) pain ≥3months and ≥3 days per week
* (2) pain intensity ≥ 40 (VAS scale from 0 no pain to 100 very painful)
* (3) the surgical indication would be based on orthopedics opinions

Exclusion Criteria:

* history of shoulder surgery in the prior 3 years
* osteoporotic vertebral fractures or rheumatologic diseases
* chronic widespread pain syndromes (fibromyalgia or chronic fatigue syndrome)
* neurological disease (i.e., stroke, parkinson's disease, etc..)
* psychiatric disease (i.e., dementia, depression, schizophrenia, etc)
* cancer
* patients who practiced yoga, meditation, chi-qong, mindfulness, or deep breathing exercises more than three times per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale change | Baseline, immediately after training, and at the 2nd, 6th, 12th, and 24th week post-operative outpatient follow-up appointments.
  Subjective post-surgical pain. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Shoulder function change_1 | Baseline, and at the 6th, 12th, and 24th week post-operative outpatient follow-up appointments.
  American Shoulder and Elbow Surgeons Shoulder Score (ASES). Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Shoulder function change_2 | Baseline, and at the 6th, 12th, and 24th week post-operative outpatient follow-up appointments.
  Constant Score to measure the objective ROM. Scores range from 0 to 100 points, representing worst and best shoulder function, respectively.
Subjective sleep quality change | Baseline, and at the 2nd, 6th, 12th, and 24th week post-operative outpatient follow-up appointments.
  Pittsburgh sleep quality index (PSQI). The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Emotion-related measurements change | Baseline, and at the 2nd, 6th, 12th, and 24th week post-operative outpatient follow-up appointments.
  Hospital Anxiety and Depression Scale (HADS) to measure anxiety and depression in the medical setting. Higher scores indicate greater anxiety and depression.
HRQoL change | Baseline, and at the 2nd, 6th, 12th, and 24th week post-operative outpatient follow-up appointments.
  EQ-5D-5L is a standardized measure of health-related quality of life. The higher transformed scores, the better HRQoL

SECONDARY OUTCOMES:
Pain-related fear | Baseline as predictive factor.
  Tampa scale of kinesiophobia. The lower TSK total scores means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia. Total scores range from 17 to 68 points.
Pain catastrophizing | Baseline as predictive factor.
  Pain catastrophizing Scale (PCS). People are asked to indicate the degree to which they have the above thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52), along with three subscale scores assessing rumination, magnification and helplessness.
Neuropsychological change - general cognitive ability | Baseline, and at the 24th week post-operative outpatient follow-up appointments.
  Montreal Cognitive Assessment (MoCA) assesses general cognitive ability. The higher scores, the better the cognitive function. The total possible score is 0~30 points; a score of 26 or above is considered normal.
Neuropsychological change - subjective cognitive ability | Baseline, and at the 24th week post-operative outpatient follow-up appointments.
  Everyday Cognition (Ecog-12) assesses subjective cognitive ability. The higher scores, the more subjective cognitive decline. The total possible score is 12~48 points; a score of 14 or above is considered as subjective decline.
Neuropsychological change - processing speed | Baseline, and at the 24th week post-operative outpatient follow-up appointments.
  Digit Symbol Coding. Under each digit the subject should write down the corresponding symbol as fast as possible. The number of correct symbols within the allowed time (e.g. 90 or 120 sec) is measured.
Neuropsychological change - working memory capacity | Baseline, and at the 24th week post-operative outpatient follow-up appointments.
  Digit span Wechsler Memory Scale III (WMS-III). The test consists of two parts forward and backward span. The participant is asked to repeat the numbers read in one second intervals in the forward span in the same order. It assesses attention, concentration and short-term memory. In the backward span, the numbers read at one-second intervals are requested to be repeated in reverse order from the end to the beginning. Working memory, which is a component of executive functions, is evaluated. The highest score that can be obtained for the forward span is 8 points, and 7 for the backward span, for a total of 15 points.
Neuropsychological change - executive control | Baseline, and at the 24th week post-operative outpatient follow-up appointments.
  Color Trails Test (CCT). The CCT is a cognitive assessment tool by connecting numbered circles and color in sequence.
HRV change | Baseline,and at the 2nd, 6th, 12th, and 24th week post-operative outpatient follow-up appointments.
  HRV refers to the variation in time intervals between consecutive heartbeats by measuring the time duration between R-waves (peak of the QRS complex) on an electrocardiogram (ECG) signal. HRV parameters could be frequency-domain, including low-frequency (LF) and high-frequency (HF) power, and time-domain, including the root mean square of successive differences (RMSSD), and the standard deviation of the IBI of normal sinus beats (SDNN).
Objective sleep parameters change | Baseline,and at the 2nd, and 24th week post-operative outpatient follow-up appointments.
  Objective sleep parameters will be measured using the wearable device and sleep diary. These sleep parameters include sleep onset latency (SOL), total sleep time (TST), sleep efficiency (SE), and wake after sleep onset (WASO).
Neurophysiological change_1 | Baseline, and at the 24th week post-operative outpatient follow-up appointments.
  Change in brain activity at rest.
Neurophysiological change_2 | Baseline, and at the 24th week post-operative outpatient follow-up appointments.
  Changes in Amplitude (μv) of EEG signals for event-related potential components.

OTHER OUTCOMES:
Cytokine | During surgery
  Joint fluid or plasma will be obtained via aspiration from the shoulder joint of each patient at the beginning of the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hao Chiu, M.D., Study Chair — Chang Gung MH
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided